CLINICAL TRIAL: NCT05840380
Title: The Effect of Graston Technique on Pain, Proprioception, Flexibility, and Disability in Patients With Chronic Non-specific Low Back Pain
Brief Title: Instrumental Soft Tissue Mobilization in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Backache
Record Dates: First submitted 2023-04-12; First posted 2023-05-03 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Low Back Pain
Keywords: Low back pain; instrumental soft tissue mobilization; flexibility; functionality; quality life
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Thirty patients (mean age; 38.46±9.03 years) with CNLBP were included in the study. The patients have randomly divided into two groups Graston technique (GT) and control. Graston was applied three times a week for four weeks in addition to the exercise program in the GT group, while only the exercise program was applied to the control group. Pain intensity (Visual analog scale), pressure pain threshold (algometer), proprioception (digital inclinometer), flexibility (sit and reach test), disability (Oswestry disability index), and quality of life (Short form-36) were evaluated at the beginning and end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise+1ASTM group (Active Comparator): In addition to the exercises given to the exercise group to the IASTM group 8-10 repetitions with the device at a 45° angle twice a week for 4 weeks on erector spines, glutes maximus, gluteus medius and hamstrings Superficial and deep fascia will be applied. Individual supine for application will be deposited. The Graston instrument glides over the tissues of the individual.
  cream will be applied to make it easier, then the physiotherapist will will stand on its side at the level and graston for 5 minutes. superficially on the thoracolumbal fascia between the sacrum and T12. will be applied. They will perform the low back pain exercises shown. Pain intensity of all patients at the beginning and end of treatment Visual Analogue Scale and algometer, flexibility sit and lie test, position sense digital inclinometer, functional status Oswestry Disability Index and life Quality will be evaluated with Short Form-36 (SF-36).
  Interventions: Device: instrumental soft tissue mobilization
- exercise group (Active Comparator): The exercise group is; By physiotherapists 3 times a week for 4 weeks They will perform the low back pain exercises shown. Pain intensity of all patients at the beginning and end of treatment Visual Analogue Scale and algometer, flexibility sit and lie test, position sense digital inclinometer, functional status Oswestry Disability Index and life Quality will be evaluated with Short Form-36 (SF-36).
  Interventions: Device: instrumental soft tissue mobilization

INTERVENTIONS:
Device: instrumental soft tissue mobilization — Individual supine for application will be deposited. The Graston instrument glides over the tissues of the individual. cream will be applied to make it easier, then the physiotherapist will will stand on its side at the level and graston for 5 minutes. superficially on the thoracolumbal fascia between the sacrum and T12. will be applied
  Other Names: exercise

SUMMARY:
Low back pain is caused by strain of the ligaments or muscles around the vertebral column or a musculoskeletal system formed due to compression of the nerves coming out of the spinal cord is a system nuisance.The process that begins as acute pain become chronic with prolongation of life, limit physical function and negatively affecting the quality of work, loss of workforce and health care It is an important health problem that causes an increase in expenditures. Thirty patients (mean age; 38.46±9.03 years) with CNLBP were included in the study. The patients have randomly divided into two groups Graston technique (GT) and control. Graston was applied three times a week for four weeks in addition to the exercise program in the GT group, while only the exercise program was applied to the control group. Pain intensity (Visual analog scale), pressure pain threshold (algometer), proprioception (digital inclinometer), flexibility (sit and reach test), disability (Oswestry disability index), and quality of life (Short form-36) were evaluated at the beginning and end of the study.This study aims to investigate the effect of the Graston technique added to exercise on pain, proprioception, disability, flexibility, and quality of life in individuals with chronic non-specific low back pain (CNLBP).

DETAILED DESCRIPTION:
Low back pain is caused by strain of the ligaments or muscles around the vertebral column or a musculoskeletal system formed due to compression of the nerves coming out of the spinal cord is a system nuisance.The process that begins as acute pain become chronic with prolongation of life, limit physical function and negatively affecting the quality of work, loss of workforce and health care It is an important health problem that causes an increase in expenditures.The most load-bearing region of the spine in the movement system is the lumbar region. from mechanical stresses, functional loads, occupational and sportive It is the area most affected by trauma. In recent years, studies have shown that manual therapy methods can be used to reduce chronic low back pain.

shows that it is a viable treatment option in reducing Instrument assisted soft tissue mobilization (Instrument Assisted Soft Tissue Mobilization, IASTM), is a popular method that can be used for myofascial restriction. is a treatment method. Reducing pain in the area of IASTM pathology, increasing range of motion (ROM), improving motion function and is used to give a mobilizing effect.In the light of studies in the literature, patients with chronic non-specific low back pain Instrumental soft tissue mobilization to be applied will reduce pain, joint range of motion, flexibility, functionality and quality of life positively is thought to develop.Thirty patients (mean age; 38.46±9.03 years) with CNLBP were included in the study. The patients have randomly divided into two groups Graston technique (GT) and control. Graston was applied three times a week for four weeks in addition to the exercise program in the GT group, while only the exercise program was applied to the control group. Pain intensity (Visual analog scale), pressure pain threshold (algometer), proprioception (digital inclinometer), flexibility (sit and reach test), disability (Oswestry disability index), and quality of life (Short form-36) were evaluated at the beginning and end of the study.This study aims to investigate the effect of the Graston technique added to exercise on pain, proprioception, disability, flexibility, and quality of life in individuals with chronic non-specific low back pain (CNLBP).

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-60
* Being diagnosed with chronic non-specific low back pain
* Volunteer to participate in the study

Exclusion Criteria:

* Psychological disorder, mental disorder, cancer and severe depression to have situations
* Primary or metastatic spinal malignancy, history of spinal fracture
* Neurological disease (Hemiplegia, Multiple Sclerosis, Parkinson, etc.)
* Having been diagnosed with advanced osteoporosis
* Surgery or acute infection of the lumbar region to be
* Patients using regular analgesics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | baseline and 4 weeks post-intervention
  Low back pain severity was measured using the Visual Analog Scale. Scale (VAS). The VAS is a 10 cm scale, where 0 represented no pain and 10 represented unbearable pain. Pain intensity was recorded by measuring the point marked between 0- 10.
Pressure pain threshold | baseline and 4 weeks post-intervention
  Pressure pain threshold (PPT) was measured using an algometer. Algometer is a device that measures sensitivity to pain caused by pressure or force applied to any part of the body. The algometer was placed vertically 2 cm lateral to the 3rd lumbar vertebra, and then the pressure was applied to the area at a rate of 1 kg/s. The point at which the patient felt an unpleasant sensation or pain was accepted as the pressure pain threshold.
Flexibility | baseline and 4 weeks post-intervention
  Sit and Reach Flexibility Test was used to evaluate trunk and hamstring muscle flexibility. Patients rested their feet on the sit-and-reach table with their knees extended. Then, they were asked to lie forward with their hands together without lifting their knees. The test was repeated 3 times and the best distance the patient reached was recorded.
Proprioception | baseline and 4 weeks post-intervention
  The sense of position, known as the sense of repositioning of the trunk, was evaluated with a digital inclinometer. The inclinometer was placed on the lumbar spinous processes while the patients stood upright. For trial and learning, they were asked to bend forward three times at 15° and 30° with their eyes closed and stop there for 3 seconds. The same procedure was applied after the trial, and the patients repeated the test 3 times. Deviation angles were recorded for 15° and 30° trunk flexion.
Disability | baseline and 4 weeks post-intervention
  The Oswestry Disability Index (ODI) was used to evaluate the level of functional disability caused by chronic low back pain [23]. The scale has ten subgroups. Subgroups of the scale: severity of pain, lifting and carrying, walking, sitting, standing, sleep, sexual life, traveling and social life. Each subgroup has six options, and the first statement is scored as "0" and the sixth statement as "5". As the total score increases, the level of disability also increases.
Quality of life-SF 36 | baseline and 4 weeks post-intervention
  The Short Form-36 (SF-36) was used to measure changes in quality of life (QoL) levels due to chronic low back pain. This scale consists of 36 items and includes physical function, physical role, bodily pain, general health, emotional role, social function, mental health, and vitality sub-parameters

CONTACTS AND LOCATIONS:
Overall Officials: Metehan YANA PhD, Principal Investigator — Karabuk Univercity
Locations (1):
- Karabük University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Moffett J, McLean S. The role of physiotherapy in the management of non-specific back pain and neck pain. Rheumatology (Oxford). 2006 Apr;45(4):371-8. doi: 10.1093/rheumatology/kei242. Epub 2005 Dec 6. PMID 16332949
- [Background] Davis KG, Marras WS. The effects of motion on trunk biomechanics. Clin Biomech (Bristol). 2000 Dec;15(10):703-17. doi: 10.1016/s0268-0033(00)00035-8. PMID 11050352
- [Background] Meier ML, Vrana A, Schweinhardt P. Low Back Pain: The Potential Contribution of Supraspinal Motor Control and Proprioception. Neuroscientist. 2019 Dec;25(6):583-596. doi: 10.1177/1073858418809074. Epub 2018 Nov 2. PMID 30387689
- [Background] Tong MH, Mousavi SJ, Kiers H, Ferreira P, Refshauge K, van Dieen J. Is There a Relationship Between Lumbar Proprioception and Low Back Pain? A Systematic Review With Meta-Analysis. Arch Phys Med Rehabil. 2017 Jan;98(1):120-136.e2. doi: 10.1016/j.apmr.2016.05.016. Epub 2016 Jun 16. PMID 27317866
- [Background] Kent P, Mjosund HL, Petersen DH. Does targeting manual therapy and/or exercise improve patient outcomes in nonspecific low back pain? A systematic review. BMC Med. 2010 Apr 8;8:22. doi: 10.1186/1741-7015-8-22. PMID 20377854
- [Background] Descarreaux M, Blouin JS, Teasdale N. Repositioning accuracy and movement parameters in low back pain subjects and healthy control subjects. Eur Spine J. 2005 Mar;14(2):185-91. doi: 10.1007/s00586-004-0833-y. Epub 2004 Nov 30. PMID 15759173
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914